CLINICAL TRIAL: NCT02298374
Title: Evaluation of Homecare Reablement, the Trondheim Model
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no funding
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: Trondheim Kommune (Other); St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2014/436
Record Dates: First submitted 2014-10-03; First posted 2014-11-24 (Estimated); Last update posted 2017-04-21 (Actual); Status verified 2017-04

CONDITIONS: Mobility Limitation; Asthenia
Keywords: Rehabilitation; Evaluation studies; Home care services
MeSH Terms: conditions — Mobility Limitation; Asthenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Homecare reablement (Experimental): Receives comprehensive assessment and individualized follow-up according to a plan with short and longterm goals.
  Interventions: Other: Homecare reablement
- Usual care (Active Comparator): Receives normal care
  Interventions: Other: usual care

INTERVENTIONS:
Other: Homecare reablement
  Arms: Homecare reablement
Other: usual care
  Arms: Usual care

SUMMARY:
The aim is to evaluate a model of home-based rehabilitation. The intervention targets elder persons who receive homecare services, but still are relatively independent in most activities of daily living. The model focuses on early identification of decline in function and intervention in the home environment through close cooperation between the participant, homecare services and therapists.

ELIGIBILITY:
Inclusion Criteria:

* receive homecare services
* live within the catchment area

Exclusion Criteria:

* In-patient length of stay (IPLOS) score > 2.0
* severe dementia

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-11; Primary Completion 2017-01 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Change in Activity level (measured by body-worn sensors) | 1 years
  measured by body-worn sensors over 4 days

SECONDARY OUTCOMES:
Change in Short Physical performance battery score | 1 year
  Performance based test of lower extremity function
Change in received hours with homecare services | 1 year
  Including nursing, assistance in activities of daily living and domestic work
Qualys (EQ- 5D) | 1 year
  EQ- 5D
Change in IPLOS score | one year
  A composite score on level of dependency in 17 different areas related to activities of daily living, including cognitive function
Change in cognitive function (Subscore of the Iplos score) | one year
  Subscore of the Iplos score

CONTACTS AND LOCATIONS:
Overall Officials: Jorunn L Helbostad, phd prof, Principal Investigator — Norwegian University of Science and Technology